CLINICAL TRIAL: NCT00030602
Title: A Phase 2 Study Of Prostate Specific Antigen-3 (PSA-3) (NSC # 694155) With Montanide (NSC #675756) Vaccination In Patients With Prostate Cancer Recurrent
Brief Title: Vaccine Therapy in Treating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MSGCC-0074; CDR0000069181 (Registry Identifier: PDQ (Physician Data Query)); NCI-2812
Record Dates: First submitted 2002-02-14; First posted 2004-02-19 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — incomplete Freund's adjuvant

INTERVENTIONS:
Biological: PSA prostate cancer vaccine
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have recurrent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of PSA-3 peptide vaccine emulsified in Montanide ISA-51 on PSA levels in patients with recurrent prostate cancer. II. Determine the toxicity of this regimen in these patients. III. Determine whether the T lymphocyte immune response to PSA-3 and HLA-A2 antigen-presenting cells that endogenously produce PSA is increased in patients treated with this regimen. IV. Determine the duration of the PSA and/or immune responses in patients treated with this regimen. V. Correlate immune and PSA responses in patients treated with this regimen. VI. Determine the efficacy of a second (boost) vaccination with this regimen in patients with a PSA or immune response.

OUTLINE: This is a multicenter study. Patients receive PSA-3 peptide vaccine emulsified in Montanide ISA-51 subcutaneously in 2 sites on days 1, 8, 15, and 22 in the absence of unacceptable toxicity. Patients who show an immune or prostate specific antigen (PSA) response are followed until disease progression, defined as a diminution or disappearance of an immune response or 2 consecutive increases in PSA over the nadir. Patients are eligible for a second series of injections at the time of progression.

PROJECTED ACCRUAL: A total of 14-44 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the prostate Previously treated with radical prostatectomy at least 3 months ago HLA-A2 positive PSA greater than 0.5 ng/mL and rising At least 0.3 ng/mL greater than post-prostatectomy nadir Confirmed by at least 2 additional PSA levels at least 2 weeks apart No bone metastases by bone scan within past 3 months No clinical evidence of local disease recurrence (no palpable mass or induration in prostatic fossa)

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 OR Karnofsky 70-100% Life expectancy: More than 1 year Hematopoietic: WBC at least 3,000/mm3 Hepatic: Bilirubin normal AST and ALT no greater than 2.5 times upper limit of normal Renal: Creatinine normal Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: Fertile patients must use effective contraception HIV negative No clinical immune dysfunction illness (e.g., rheumatoid arthritis) No ongoing or active infection No other concurrent uncontrolled illness that would preclude study No concurrent psychiatric illness or social situation that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Neoadjuvant hormonal therapy prior to prostatectomy allowed No concurrent hormonal therapy for recurrent prostate cancer Radiotherapy: No prior radiotherapy to the prostate No prior radiotherapy to the pelvis Surgery: See Disease Characteristics Other: No other concurrent investigational agents No concurrent commercial agents intended to treat the malignancy No concurrent immunosuppressive therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01 (Actual); Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Dawson, MD, Study Chair — University of Maryland Greenebaum Cancer Center